CLINICAL TRIAL: NCT04229446
Title: In What Way do Music-based Caregiving Influence Pain, Daily Activity, QOL, Neuropsychiatric Symptoms, and Medication in Patients With Dementia
Brief Title: Music Based Caregiving in Patients With Pain and Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Helse Midt-Norge (Other); St. Olavs Hospital (Other); University of Oslo (Other); University of Bergen (Other); Norwegian Centre for Ageing and Health (Other)
Responsible Party: Principal Investigator, Tone Rustøen, Professor, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2018/2519
Record Dates: First submitted 2019-10-09; First posted 2020-01-18 (Actual); Results first posted 2023-12-07 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-02

CONDITIONS: Pain; Dementia; Music; Activity, Motor; Quality of Life
MeSH Terms: conditions — Pain; Dementia; Motor Activity

STUDY DESIGN:
Intervention Model Description: This is a cluster-randomized controlled trial including patients with dementia and pain living at different wards at nursing homes.
Who Masked: Outcomes Assessor
Masking Description: The included statistician will do the first evaluation of the results
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Receive the music based intervention (Experimental): After the healthcare workers have accomplished the MBC program the eight week intervention program will be applied by the trained staff at the intervention wards. The intervention (MBC) consists of daily individualized prerecorded music integrated with activity with about 30 minutes duration, combined with a one hour active session in groups twice weekly. The music will be selected based on individualized preferences from the patients or their family. The music will also be adapted to the day rhythm; awakening in the morning, support activities during the day, or for sleep in the evening. The healthcare worker will bring playback equipment e.g. a CD-player to the patient room. In addition will two weekly sessions in groups be performed (each on one hour) with music and movement. The movement will be adapted to their physical capacity.
  Interventions: Behavioral: Music based caregiving
- Standard care group (No Intervention): Standard care for participants in this group

INTERVENTIONS:
Behavioral: Music based caregiving — The intervention (MBC) consists of daily individualized prerecorded music integrated with activity with about 30 minutes duration, combined with a one hour active session in groups twice weekly. The music will be selected based on individualized preferences from the patients or their family. The music will also be adapted to the day rhythm; awakening in the morning, support activities during the day, or for sleep in the evening. The healthcare worker will bring playback equipment e.g. a CD-player to the patient room. In addition will two weekly sessions in groups be performed (each on one hour) with music and movement.
  Arms: Receive the music based intervention

SUMMARY:
The main objective of this study is to evaluate the pain-relieving effect of a well-characterized non-pharmacological treatment program, music-based caregiving (MBC), to patients in nursing homes with dementia and pain. Patients with dementia disease will be recruited from nursing homes in Trondheim and Oslo, and each ward at the nursing homes will be cluster randomized into intervention - or control wards. Then the health care personnel in the intervention wards will receive education in MBC and perform the intervention during eight weeks. The hypothesis is that this non-pharmacological intervention will reduce pain intensity and improve general activity, as well as reduce other symptoms in nursing home patients with dementia and pain compared to baseline.

DETAILED DESCRIPTION:
This is a cluster-randomized controlled trial including patients with dementia and pain living at different wards at eight nursing homes.

1. About 12 nursing homes are selected to participate in Trondheim and in Oslo.
2. All patients at the included nursing homes will be screened with respect to dementia and pain (see screening tools later). If patients have dementia and report pain (≥3 on MOBID 2) they will be included in the intervention part of the study (n=240).
3. The included patients will then have a clinical examination of pain and pain management by expert physicians (see below). Evaluation of the use of analgesics and psychopharmacological medication will be performed. Inappropriate medication (both too much and too little) will be corrected in collaboration with the nursing home doctor.
4. In addition to the clinical examination of pain, the investigators will measure total daily physical activity, ADL, QOL, and neuropsychiatric symptoms on all included patients.
5. After the pre-test - a randomization of the wards into intervention wards or control wards will be performed.
6. About five staff members at each of the wards randomized to the intervention group will receive education in the MBC before intervention.
7. A post-test just after the intervention has ended, pain, total daily physical activity, ADL, QOL, and neuropsychiatric symptoms will be measured.

ELIGIBILITY:
Inclusion Criteria:

* All patients living in one of the included nursing homes in Oslo or Trondheim will be included in the first descriptive phase
* Patients will be included in the intervention part if they report moderate pain or more (≥3 on MOBID) and mild dementia or more (≥1 on CDR).

Exclusion Criteria:

* They will not be included if they have lived in the nursing home less than four weeks, have short (less than eight weeks) expected lifetime (judged by the nurses),or if they do not understand the Norwegian language.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2020-08-05 (Actual); Study Completion 2020-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tone Rustøen, PhD, Principal Investigator — Oslo University Hospital
Locations (2):
- Norway (2):
  - Oslo University Hospital, Oslo
  - St. Olavs hospital Trondheim University Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Myrenget ME, Rustoen T, Myskja A, Smastuen M, Rangul V, Hapnes O, Borchgrevink PC, Butler S, Selbaek G, Husebo B, Sandvik R. The effect of a music-based caregiving intervention on pain intensity in nursing home patients with dementia: a cluster-randomized controlled study. Pain. 2024 Jul 1;165(7):1550-1558. doi: 10.1097/j.pain.0000000000003156. Epub 2024 Jan 2. PMID 38189182
- [Derived] Myrenget ME, Borchgrevink PC, Rustoen T, Butler S, Thorsvik D, Smastuen MC, Sandvik R. Chronic pain conditions and use of analgesics among nursing home patients with dementia. Pain. 2023 May 1;164(5):1002-1011. doi: 10.1097/j.pain.0000000000002794. Epub 2022 Dec 21. PMID 36542760

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Care Group: The participants allocated to this group received the best of standard care.
Period: Overall Study
Arm/Group | Receive the Music Based Intervention | Standard Care Group
Started | 134 | 142
Completed | 117 | 124
Not Completed | 17 | 18
Not completed — Death | 12 | 10
Not completed — Lost to Follow-up | 5 | 8

BASELINE CHARACTERISTICS:
Population: Screening: 330 in the intervention and 317 in the standard care group For pretest (baseline) we included 134 in the intervention group and 142 in the standard care.
Groups:
- Standard Care Group: The patients will receive thei best of stand care
- Total: Total of all reporting groups
Arm/Group | Receive the Music Based Intervention | Standard Care Group | Total
Number analyzed (Participants) | 134 | 142 | 276
Age, Categorical [Count of Participants; unit: Participants] — These are the participants in the screening where we included the birth date and enrolment date to calculate age.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 1 | 1 | 2
    >=65 years | 133 | 141 | 274
Age, Continuous [Mean (Full Range); unit: years] — We collected the birth date of the included participant and used the date of enrolment to calculate the age.
  years | 87 [59 to 102] | 86 [55 to 103] | 86 [55 to 103]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 100 | 196
  Male | 38 | 42 | 80
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Norway | 134 | 142 | 276
MOBID-2 pain scale [Mean (Full Range); unit: units on a scale] | 5 [0 to 10] | 5 [0 to 10] | 5 [0 to 10]

OUTCOME MEASURES:

1. Primary Outcome: Pain Occurence
Description: MOBID 2 observation instrument. The assessment of inferred pain intensity is observed based on patient's pain behaviors during standardized, guided movements of different body parts (Part 1). In addition, MOBID-2 includes an observation of pain behavior related to internal organs, head and skin registered on pain drawings and monitored over time (Part 2). MOBID-2 has shown to be reliable, valid and time-effective to assess pain in patients with severe dementia. The investigators will use MOBID-2 for assessment of pain in all the patients with dementia. Scoring range is 0-10, the higher the score the more pain.
Time Frame: 8 weeks
Measure: Mean (95% Confidence Interval); unit: units on Mobid-2 pain scale ( 0-10)
Groups:
- Standard Care Group: Standard care will be provided
Arm/Group | Receive the Music Based Intervention | Standard Care Group
Number analyzed (Participants) | 134 | 142
units on Mobid-2 pain scale ( 0-10) | 4.6 [4.3 to 4.8] | 4.6 [4.4 to 4.8]

2. Secondary Outcome: The Total Daily Physical Activity
Description: Two three-axis accelerometers attached to the skin on the right thigh and low back for seven continuous days. By utilizing state-of-the-art machine-learning techniques, the investigators have developed a preliminary activity recognition model for lying, sitting, standing, walking and other activities. This model has been used in the Nord-Trøndelag health study (HUNT4). Specifically, the model captures walking velocity and transitions between postures and activities (e.g. sit-to-stand) and sleep quality/duration.
Time Frame: 8 weeks
Reporting Status: Not Posted, anticipated posting 2024-12

3. Secondary Outcome: Stage of Dementia Disease
Description: Clinical Dementia Rating Scale (CDR) is an assessment scale for the accurate clinical staging of dementia in older subjects. The CDR includes six items assessing cognitive and functional impairment. Based on an algorithm giving precedence to the item memory a total score is estimated. A score of 0, 0.5, 1, 2, 3 indicates no dementia, questionable dementia, mild, moderate or severe dementia, respectively, and CDR score > 1, is cut-off score for dementia disease. The scale has shown to be reliable and valid, also the Norwegian version.
Time Frame: 8 weeks
Reporting Status: Not Posted, anticipated posting 2024-12

4. Secondary Outcome: Neuropsychiatric Symptoms
Description: The Neuropsychiatric Inventory (NPI-NH) measure 12 different psychiatric symptoms and behavioural disturbances in nursing home residents: delusions, hallucinations, dysphoria, anxiety, agitation/aggression, euphoria, disinhibition, irritability/lability, apathy, aberrant motor activity, sleep and night-time behaviour disorders, appetite and eating disorders. The screening question is asked to determine if the behavioural change is present. If a screening question is present, there will be sub-questions about frequency (score 1 to 4) and intensity (score 1 to 3) for each behavior. Total score for each behavior is from 1 to 12. The total scoring range is from 0-144, the higher the score the more symptoms. The scale has been validated for patients in nursing homes in Norway.
Time Frame: 8 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Depression
Description: Cornell scale for depression in dementia assesses signs and symptoms of major depression in patients with dementia in an interview with the health care providers. The scale consists of 19 items in five domains based on observation of behaviour. Each question is scored on a two-point scale: 0=absent; 1=mild or intermittent; 2=severe; n/a = unable to evaluate.
Time Frame: 8 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Level of Quality of Life: QUALID-scale
Description: Quality of Life in Late-Stage Dementia (QUALID) measures QOL in patients with severe dementia based on information and observations from nurses about the patient's emotions and behavior. Dementia Quality of Life (DQoL) will also be used as QUALID-scale is an observation scale, and there is a lack of studies comparing self-reported and observations QoL in those with dementia, the investigators want to compare the observation estimate with self-report for patients with none, mild and moderate dementia (DQoL). DQoL consists of five domains: self-esteem, positive affect/ humor, feeling of belonging, and sense of aesthetics and negative affect. The instrument is evaluated in those with mild and moderate dementia and is used in nursing homes in Norway. Scoring range is from 11-55, the higher the score the worse QOL.
Time Frame: 8 weeks
Reporting Status: Not Posted, anticipated posting 2024-12

7. Secondary Outcome: Aids of Daily Living
Description: Barthel's Activities of Daily Living Index (ADL) is a screening instrument for patients' daily life functioning. This 10-point scale measures patients' degree of self-reliance with a total score ranging from 0 to 20. Lower scores indicate greater dependence on nursing care.
Time Frame: 8 weeks
Reporting Status: Not Posted, anticipated posting 2024-12

ADVERSE EVENTS:
Time Frame: We monitored effects and side-effects during the intervention period of eight (8) weeks.
Description: we used the definitions as described.
Groups:
- Standard Care Group: Standard care. Participants receive their care as usual.
Arm/Group | Receive the Music Based Intervention | Standard Care Group
All-Cause Mortality (participants affected / at risk) | 12/134 | 10/142
Serious Adverse Events (participants affected / at risk) | 0/134 | 0/142
Other Adverse Events (participants affected / at risk) | 0/134 | 0/142

LIMITATIONS AND CAVEATS:
-Possible selection bias

1. Patients selected from 12 different nursing homes in 2 different cities in Norway using different selection strategies. In Oslo, an invitation email was sent to all nursing homes, and the ones interested responded, whereas in Trondheim, the nursing homes were chosen by the municipality.
2. Our study does not include nursing homes from rural areas and thus may not be truly representative for the general nursing home population in Norway

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-25): https://cdn.clinicaltrials.gov/large-docs/46/NCT04229446/Prot_SAP_000.pdf